CLINICAL TRIAL: NCT05699655
Title: Tislelizumab Combined With Apatinib and Oxaliplatin Plus S1 Vs Oxaliplatin Plus S1 as Neoadjuvant Therapy for Borrmann IV、Large Borrmann III Type and Bulky N Positive Advanced Gastric Cancer: Randomized Control, Open, Multicenter Trial-2 (TAOS-3B-Trial-2)
Brief Title: Tislelizumab Combined With Apatinib and Oxaliplatin Plus S1 Vs Oxaliplatin Plus S1 as Neoadjuvant Therapy for Borrmann IV、Large Borrmann III Type and Bulky N Positive Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAOS-3B Trial 2
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-05

CONDITIONS: Immunotherapy Gastrict Cancer
MeSH Terms: interventions — tislelizumab; apatinib; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with apatinib and oxaliplatin plus S1 (Experimental)
  Interventions: Drug: Tislelizumab; Drug: apatinib; Drug: oxaliplatin; Drug: S-1
- oxaliplatin plus S1 (Active Comparator)
  Interventions: Drug: oxaliplatin; Drug: S-1

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks for 4 cycles. Discontinuation will be considered due to toxicity, withdrawal of consent, or end of study. Every 3-week treatment period was considered to be a cycle.
  Arms: Tislelizumab combined with apatinib and oxaliplatin plus S1
Drug: apatinib — Participants will receive apatinib, 250mg, qd，every 3 weeks for 3 weeks
  Arms: Tislelizumab combined with apatinib and oxaliplatin plus S1
Drug: oxaliplatin — Participants will receive oxaliplatin, 130mg/m2, day 1 of every 3 weeks for 4 weeks.
Drug: S-1 — Participants will receive S-1, day 1-14 of every 3 weeks for 4 weeks.

SUMMARY:
To evaluate the clinical efficacy and safety of Tislelizumab combined with apatinib mesylate, oxaliplatin plus S1 Vs oxaliplatin plus S1.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years of age.
* Histologically confirmed gastric adenocarcinoma was diagnosed in patients with locally advanced gastric cancer with tumor volume >5cm Borrmann III, Borrmann IV and BulkyN according to AJCC Version 8.
* Measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.
* ECOG（Eastern Cooperative Oncology Group）PS（Performance Status）:0-1 scores.
* No previous surgical treatment, anti-tumor chemoradiotherapy/immunotherapy was performed.
* Preoperative endoscopic examination confirmed no positive peritoneal implantation metastasis and exfoliated cells.
* The expected survival time is more than 6 months.
* For women of reproductive age, a urine or serum pregnancy test with negative results should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1).If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested.Women of childbearing age were defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy.

Exclusion Criteria:

* Diagnosis of malignant diseases other than gastric cancer within 5 years prior to first administration (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or radical resectable carcinoma in situ).
* Significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis, etc. occurred within 3 months before enrollment. If fecal occult blood was positive at baseline, reexamination could be performed，if it was still positive after reexamination, gastroscopy was required.
* Prior treatment: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T-cell receptor (e.g., CTLA-4, OX-40, CD137).
* A history of immunodeficiency, including HIV testing positive.
* Is currently participating in an interventional clinical study or has been treated with another study drug or study device in the 4 weeks prior to initial dosing.
* Patients who had a history of cardiovascular and cerebrovascular diseases and were still taking thrombolytic drugs or anticoagulants orally.
* HER2 positive is known.
* Patients with previous gastrointestinal perforation, abdominal abscess or recent intestinal obstruction (within 3 months) or imaging or clinical symptoms suggesting intestinal obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 4 weeks after surgery
  Total tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Major pathological response | 4 weeks after surgery
  Total/moderate tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Objective Response Rate (ORR) | At the end of Cycle 3 (each cycle is 21 days)]
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China